CLINICAL TRIAL: NCT01584453
Title: A Randomised, Double-blind, Placebo-controlled Trial Assessing the Safety and Efficacy of Intracoronary Nitrite Infusion During Acute Myocardial Infarction
Brief Title: Safety and Effectiveness of Intra-coronary Nitrite in Acute Myocardial Infarction
Acronym: NITRITE-AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/LO/1500
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2015-07

CONDITIONS: Myocardial Infarction; Reperfusion Injury; Myocardial Ischemia; Cardiovascular Diseases
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury; Myocardial Ischemia; Cardiovascular Diseases | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Nitrite (Experimental)
  Interventions: Drug: Sodium Nitrite
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium Chloride Placebo

INTERVENTIONS:
Drug: Sodium Nitrite — A bolus of sodium nitrite solution (1.8 micromol in 10 ml PRe-diluted in 0.9% sodium chloride in a syringe) will be delivered over 30-60 seconds via intracoronary injection initiated during the re-establishment of antegrade epicardial flow with PPCI.
  Arms: Sodium Nitrite
Drug: Sodium Chloride Placebo — The control intervention is a bolus of 0.9% sodium chloride solution (prepared with an identical appearance to the sodium nitrite).
  Arms: Placebo

SUMMARY:
Despite advances in the treatment of heart attacks the complications and death rates from failure of the heart to pump properly after treatment remain high. A heart attack occurs when one or more of the arteries that supply blood to the heart become blocked, causing the heart to be starved of oxygen and nutrients. This results in damage to the heart and so the the heart pumps less well. The main treatment for a heart attack is balloon treatment to open the blocked artery (called primary angioplasty). Whilst re-opening the artery is essential and allows blood to flow to the area of the heart starved of oxygen, this process also causes damage itself (called reperfusion injury) and increases the size of the heart attack further. Currently there are no treatments available that reduce this reperfusion injury. The investigators and others have shown that a substance called sodium nitrite reduces reperfusion injury in experimental models of a heart attack. The aim of this research is to perform a trial to investigate whether during a heart attack, an infusion of sodium nitrite into the damaged artery protects against reperfusion injury and reduces heart attack size in patients.

DETAILED DESCRIPTION:
Coronary heart disease is still the commonest cause of death in the UK (in the main as a consequence of acute myocardial infarction (AMI)). Presently, timely and effective reperfusion with primary percutaneous coronary intervention (PPCI) remains the most effective treatment strategy for limiting infarct size, preserving left ventricular ejection fraction (LVEF), and improving the clinical outcomes in such patients. However, substantial mortality and morbidity rates still persist with respect to longer term outcome. One of the main determinants of prognosis after AMI is the size of the infarct. Thus, identification of additional strategies that might decrease infarct size is desirable.

Evidence from pre-clinical studies suggests that inorganic nitrite administration reduces infarct size in animal models of AMI. In this study we aim to translate these findings into man. We will test the hypothesis that in patients with STEMI undergoing PPCI, an intra-coronary injection of nitrite, initiated prior to establishment of full reperfusion reduces infarct size through prevention of ischemia-reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years
* Acute STEMI with ECG showing ST-segment elevation of 1mm or more in two adjacent limb leads or 2mm or more in at least two contiguous precordial leads or new left bundle branch block;
* Haemodynamically stable
* Estimated symptom to balloon or aspiration time < 6 hours
* Angiographically i) PPCI indicated for revascularisation ii) Single epicardial artery to be treated iii) Expected ability to use over the wire balloon

Exclusion Criteria:

* Patients on organic nitrate treatment (Nicorandil, isosorbide mononitrate)
* Previous history of AMI, systolic dysfunction or CABG
* Subjects presenting with cardiogenic shock (systolic blood pressure <80 mmHg for > 30 minutes, or requiring inotropes/emergency intra aortic balloon pump or cardiopulmonary resuscitation
* Current diagnosis of or treatment for malignancy, other than non-melanoma skin cancer.
* Current life-threatening condition other than vascular disease that may prevent a subject completing the study.
* Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication.
* Patients considered unsuitable to participate by the research team (e.g., due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study-related procedures).
* Severe acute infection, or significant trauma (burns, fractures).
* Pregnancy.
* Contra-indications to CMR scanning i) Pacemakers, intracranial clips or other metal implants ii) Claustrophobia iii) Renal failure (eGFR < 30mls/min)
* History of alcohol or drug abuse within the past 6 months.
* History of congenital methaemoglobinaemia.
* Angiographically severe vessel tortuosity, diffuse disease or severe calcification which may impede successful delivery of the the over the wire balloon.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Infarct size measured by CK area under the curve | 1st 48 hours after AMI
  AUC measured over the 1st 48 hours after PPCI (0,4,8,12,18,24,36 and 48 hours)

SECONDARY OUTCOMES:
Infarct size measured by Troponin T Area under the curve | 1st 48 hours post AMI
  AUC measured over the 1st 48 hours after PPCI (0,4,8,12,18,24,36 and 48 hours)
Infarct size, assessed by CMR at 6 months ± 2 weeks. | 6 months ± 2 weeks.
  Infarct size, assessed by CMR at 6 months ± 2 weeks.
Infarct size as a proportion of area at risk measured at 48 hours by CMR. | 48 hours
  Infarct size as a proportion of area at risk measured at 48 hours by CMR.
The acute safety and tolerability of intra-coronary nitrite in STEMI | 1st 48 hours
  Safety profile of IC nitrate (death, MI, CVA, arrhythmia, hypotension, methaemoglobinaemia)
Assessment of MACE endpoints at 6 and 12 months (death, heart failure, myocardial infarction, stroke, need for repeat revascularisation) | 12 months
Markers of inflammation measured at baseline, 30 minutes, 4 and 24 hours post PCI | 24 hours
  hs-CRP, MCP-1
Assessment of platelet reactivity at baseline, 30 minutes, 4 and 24 hours post PCI | 24 hours
  ADP, collagen, PBS
Plasma nitrite and cyclic guanosine monophosphatase (cGMP) concentrations measured at baseline, post procedure, at 4 hours and 24 hours post-PCI | 24 hours
Cost-utility of Nitrite over at 3 years | 3 years
  ICER based on outcome and QoL (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, FRCP, PhD, Principal Investigator — Barts and the London NHS Trust/QMUL
Locations (1):
- London Chest Hospital, Bethnal Green, London, United Kingdom

REFERENCES:
- [Derived] Jones DA, Khambata RS, Andiapen M, Rathod KS, Mathur A, Ahluwalia A. Intracoronary nitrite suppresses the inflammatory response following primary percutaneous coronary intervention. Heart. 2017 Apr;103(7):508-516. doi: 10.1136/heartjnl-2016-309748. Epub 2016 Sep 28. PMID 27683405
- [Derived] Jones DA, Pellaton C, Velmurugan S, Rathod KS, Andiapen M, Antoniou S, van Eijl S, Webb AJ, Westwood MA, Parmar MK, Mathur A, Ahluwalia A. Randomized phase 2 trial of intracoronary nitrite during acute myocardial infarction. Circ Res. 2015 Jan 30;116(3):437-47. doi: 10.1161/CIRCRESAHA.116.305082. Epub 2014 Dec 15. PMID 25512434
- [Derived] Jones DA, Andiapen M, Van-Eijl TJ, Webb AJ, Antoniou S, Schilling RJ, Ahluwalia A, Mathur A. The safety and efficacy of intracoronary nitrite infusion during acute myocardial infarction (NITRITE-AMI): study protocol of a randomised controlled trial. BMJ Open. 2013 Apr 2;3(4):e002813. doi: 10.1136/bmjopen-2013-002813. Print 2013. PMID 23550096